CLINICAL TRIAL: NCT05132153
Title: Effect of Nebulized Milrinone on Right Ventricular Hemodynamics in Adult Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, samar mohammed, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAMSU R 174/2021
Record Dates: First submitted 2021-10-22; First posted 2021-11-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Milrinone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group A) will receive milrinone (Active Comparator): Patients will receive milrinone 50 microgram/kg in 5ml volume, over 5 min by nebulization
  Interventions: Drug: Milrinone
- (Group B) will receive normal saline (Placebo Comparator): Patients will receive 5 ml saline by nebulization over 5 min
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Milrinone — will be given by nebulization
  Arms: (Group A) will receive milrinone
Drug: Normal saline — will be given by nebuliztion
  Arms: (Group B) will receive normal saline

SUMMARY:
The primary aim of this study was to investigate the effect inhaled milrinone given before CPB on improving the right ventricular function measured by transesophageal echocardiography (TEE) at time of CPB separation.

DETAILED DESCRIPTION:
The investigator will include (70) patients planned for elective adult cardiac surgery (Coronary revascularization surgery, Mitral valve surgery, Aortic valve surgery or complex surgery (either two or more valves or valves and coronary revascularization surgery). All surgery should be with CPB. All patients will be diagnosed with preoperative PH. After separation of CPB the patients evaluated as regard the hemodynamics (MAP, HR), the inotropic score as additional intravenous milrinone in the case of low cardiac output or presence of post-CPB PH or RV failure with reduced contractility documented using TEE. Left ventricular EF, and right ventricular hemodynamics represented by RV function measured by (tricuspid annulus plane systolic excursion (TAPSE), fractional area change FAC), and right ventricular systolic pressure by doppler (RVSP) which represent the pulmonary artery pressure all data will be assessed by transesophageal ECHO after anesthesia, immediately before CPB and immediately after separation from CPB all these data will be recorded in the study.

ELIGIBILITY:
Eligibility criteria:

* elective adult cardiac surgery (Coronary revascularization surgery, Mitral valve surgery, Aortic valve surgery or complex surgery (either two or more valves or valves and coronary revascularization surgery).
* All surgery should be with CPB.
* All patients will be diagnosed with preoperative PH. PH was defined as a mean pulmonary artery pressure (MPAP) 30 mmHg or a systolic pulmonary artery pressure (SPAP) 40 mmHg, measured during preoperative right-sided catheterization or estimated by using doppler transthoracic echocardiography.

Exclusion Criteria:

* Cardiac surgery without CPB.
* Hemodynamic instability in the preoperative time (defined as acute requirement for vasoactive support or mechanical device).
* Adult congenital heart disease planned for corrective surgery.
* Contraindication to transesophageal echocardiography (TEE).
* Any surgery involves tricuspid valve annulus as it will compromise the accuracy of RV function assessment by TEE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-17 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Effect of inhaled milrinone on improvement of right ventricular function | After 15 minutes of inhaled milrinone intraoperative and repeated after 12, 24 hours in intensive care unit
  The right ventricle function will be assessed by Fractional area change ( Change in area between systole and diastole by echocardiograph ( intraoperative and postoperative)

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Soliman, Cairo, Nasr City, Egypt